CLINICAL TRIAL: NCT03970005
Title: Evaluation of Step-Based Care for Individuals at Clinical High Risk for Psychosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas Breitborde, Associate Professor, Ohio State University
Other Study IDs: 2018H0503
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Prodromal Schizophrenia
Keywords: psychosis; treatment; clinical high-risk
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Step-Based Care Model — Care model comprised of psychosocial and pharmacological interventions in which individuals start with low-intensity interventions and progress onto progressively higher-intensity interventions until their reach remission criteria.

SUMMARY:
The Ohio State University Early Psychosis Intervention Center is implementing a specialized clinical program to serve individuals who meet clinical high risk criteria for a psychosis. The purpose of this study is to evaluate the long-term outcomes among individuals participating in this clinical service.

DETAILED DESCRIPTION:
The Ohio State University Early Psychosis Intervention Center (OSU EPICENTER) is implementing a specialized clinical program to serve individuals ages 12-25 who meet clinical high risk criteria for a psychosis (CHR-P). The purpose of this project is to evaluate (i) correlates of baseline characteristics among clinic participants; (ii) outcomes among individuals participating in this clinical service; and (iii) predictors and mediators of longitudinal outcomes among individuals participating in this clinical service.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages 12-25
* Individuals meeting clinical high-risk criteria for psychosis as determined using the Structured Interview for Psychosis Risk. Inclusive of individuals meeting any of the three CHR syndromes assessed by the SIPS (i.e., attenuated psychotic symptoms; brief intermittent psychosis, and genetic risk and functional deterioration) and/or individuals at all four current status specifiers for the SIPS (i.e., progression, persistence, partial remission, and full remission) given evidence that future worsening of symptoms and/or progression to psychosis is possible for individuals in each current status specifier category.
* Subjects with no evidence of a pre-existing intellectual disability defined as a premorbid IQ >70 as estimated using the Reading subtest of the Wide Range Achievement Test-4
* Fluent in English per self-report

Ages: 12 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: This program evaluation will include all patients referred to The OSU EPICENTER CHR-P clinical program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Time to remission of clinical-high risk status for psychosis | Remission status assessed at all treatment visits which will occur approximately once every week for up to 104 weeks
  Using criteria inspired by Nelson et al. (2018), remission of clinical high risk status for psychosis is defined as simultaneous remission of both (i) symptoms and (ii) functional deficits associated with prodromal psychosis.
  Remission of symptoms is defined as all positive symptom items scored less than 3 on the Structured Clinical Interview for Prodromal States (SIPS). Each item is rated from 0-6 with higher scores indicating greater severity of symptoms.
  Remission of functional deficits is defined as a 5-point increase on the Personal and Social Performance scale (PSP: Morosini et al., 2000) as compared to baseline assessment or the PSP score ≥ 70. Scores range from 0-100 with higher scores indicative of better personal and social functioning.

SECONDARY OUTCOMES:
Change from baseline in quality of life assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on WHO Quality of Life Scale Brief (WHOQOL-BREF) as compared to baseline assessment
  The WHOQOL-BREF provides scores for four subscales of quality of life: physical health, psychological health, social relationships, and environment. Scores range from 0-100 with higher scores indicative of greater quality of life
Change in from baseline in cognitive functioning assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the MATRICS Consensus Cognitive Battery (MCCB) as compared to baseline assessment. The MCCB provides an overall cognitive composite score as well as subscale scores for processing speed, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem-solving, and social cognition. Scores range from 0-100 with higher scores indicative of greater cognitive functioning
Change from baseline in suicidality assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Columbia Suicide Severity Rating Scale (C-SSRS)as compared to baseline assessment. The C-SSRS provide two subscales: suicidal ideation and suicidal behavior. The former is an ordinal rating scale ranging from 0-6 with higher scores indicative of greater suicidal ideation. The latter is a nominal scale identifying the absence/presence of different suicidal behaviors.
Change from baseline in substance use severity assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the HABITS scale as compare to baseline as compared to baseline assessment. The HABITS assesses the frequency/amount of use of different illicit substances with higher scores indicative of greater frequency/amount. There is no predetermined possible range of scores as scores are raw values with regard to frequency/amount of use (e.g., number of cigarettes smoked per day)
Change from baseline in anxiety assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Hamilton Anxiety Scale scale as compared to baseline assessment.. The total score on this measure ranges from 0-56 with higher scores indicative of worse anxiety
Change from baseline in depressed mood assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Calgary Depression Scale for Schizophrenia as compared to baseline assessment. Total scores range from 0-3 with higher scores indicative of worse depression
Change from baseline in symptomatology assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Structured Interview for Psychosis Risk Syndromes as compared to baseline assessment. Item scores range from 0-6 with higher scores indicative of worse symptomatology
Change from baseline in social functioning assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Global Functioning: Social as compared to baseline assessment. Scores range from 1-10 with higher scores indicative of better social functioning
Change from baseline in role functioning assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in scores on the Global Functioning: Role as compared to baseline assessment. Scores range from 1-10 with higher scores indicative of better role functioning
Change from baseline in service utilization assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in utilization of health care and related social services as tracked using the Service Utilization and Resources Form as compared to baseline assessment.
Change from baseline in medication adherence assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in medication adherence as tracked using the Medication Adherence rating Scale as compared to baseline assessment. Scores range from 0-10 with higher scores indicative of greater adherence to prescribed medication.
Change from baseline in experience of trauma assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in experience of trauma as tracked using the Brief Trauma Questionnaire as compared to baseline assessment.
Change from baseline in health-related quality of life assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in health-related quality of life as assessed using the RAND 36-Item Health Survey as compared to baseline assessment. Scores on this measure range from 0-100 with higher scores indicative of greater health-related quality of life.

OTHER OUTCOMES:
Change from baseline in capability for suicide/lethal self-injury assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in capability for suicide/lethal self-injury as assessed using the Acquired Capacity for Suicide Scale as compared to baseline assessment. Higher scores on this measure are indicative of greater capability for suicide/lethal self-injury.
Change from baseline in beliefs about use of alcohol assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in belief about use of alcohol as assessed using the Alcohol Expectancy Questionnaire as compared to baseline assessment. Higher scores on this measure are indicative of more positive beliefs about use of alcohol
Change from baseline in beliefs about use of marijuana assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in belief about use of alcohol as assessed using the Marijuana Effect Expectancy Questionnaire as compared to baseline assessment. Higher scores on this measure are indicative of more positive beliefs about use of marijuana
Change from baseline in recognition of predilection to common thinking errors assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in recognition of predilection to common thinking errors as assessed using the Beck Cognitive Insight Scale as compared to baseline assessment. Higher scores on this measure are indicative of greater recognition of one's predilection to common thinking errors
Change from baseline in perceptions of core qualities of self and others assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in perception of core qualities of self and others as assessed using the Brief Core Schema Scale as compared to baseline assessment. Scores on this measure assess whether an individual maintains more positive or negative perceptions about themselves and other people
Change from baseline in cognitive biases commonly experienced by individuals with psychosis assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in cognitive biases commonly experienced by individuals with psychosis as assessed using the Cognitive Biases Questionnaire in Psychosis as compared to baseline assessment. Scores on this measure assess whether an individual is more likely to experience cognitive biases commonly experienced by individuals with psychosis
Change from baseline in executive functioning assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in executive functioning as assessed using the Delis-Kaplan Executive Functioning System as compared to baseline assessment. Higher scores on this measure are indicative of greater executive functioning skills.
Change from baseline in motor functioning assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in motor functioning as assessed using the Finger Tapping Test and Grooved Pegboard as compared to baseline assessment. Higher scores on these measures are indicative of greater motor functioning.
Change from baseline in Body Mass Index (BMI) as assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in BMI as compared to baseline assessment. BMI to be calculated as kg/m^2
Change from baseline in resting blood pressure as assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in resting blood pressure as compared to baseline assessment.
Change from baseline in resting pulse as assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in resting pulse as compared to baseline assessment.
Change from baseline in theory of mind assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in theory of mind as assessed using the Hinting Task and the Movie for the Assessment of Social Cognition as compared to baseline assessment. Higher scores on these measures are indicative of greater theory of mind.
Change from baseline in internalized stigma associated with a mental illness assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in internalized stigma as assessed using the Internalized Stigma of Mental Health Scale as compared to baseline assessment. Higher scores on this measures are indicative of greater internalized stigma.
Change from baseline in experienced stigma associated with a mental illness assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in experienced stigma as assessed using the Stigma Questionnaire as compared to baseline assessment. Higher scores on this measures are indicative of greater experience of stigma.
Change from baseline in level of physical activity assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in level of physical activity assessed using the International Physical Activity Questionnaire as compared to baseline assessment. Higher scores on this measures are indicative of greater level of physical activity.
Change from baseline in perceived belongingness and perceived burdensomeness assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in perceived belongingness and perceived burdensomeness assessed using the Interpersonal Needs Questionnaire as compared to baseline assessment. Higher scores on this measures are indicative of lower perceived belongingness and greater perceived burdensomeness.
Change from baseline in insight into cognitive abilities assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in insight into cognitive abilities assessed using the Measure of Insight into Cognition as compared to baseline assessment. Higher scores on this measures are indicative of greater insight into cognitive abilities.
Change from baseline in metacognition assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in metacognition assessed using the Metacognition Awareness Inventory and modified Zoo Task as compared to baseline assessment. Higher scores on these measures are indicative of greater metacognitive abilities.
Change from baseline in use of tobacco products assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in use of tobacco products assessed using the PATH Assessment of Tobacco Use as compared to baseline assessment. This measure track rate of use of different tobacco products
Change from baseline in symptomatology associated with Post Traumatic Stress Disorder assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in symptomatology associated with Post Traumatic Stress Disorder assessed using the PTSD Checklist-5 as compared to baseline assessment. Higher scores on this measure are associated with greater severity of symptoms associated with PTSD
Change from baseline in quality of socialization assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in quality of socialization assessed using the Quality of Socialization Questionnaire as compared to baseline assessment. Higher scores on this measure are associated with greater quality of socialization
Change from baseline in referential thinking assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in referential thinking assessed using the Referential Thinking Scale as compared to baseline assessment. Higher scores on this measure are associated with greater referential thinking
Change from baseline in perceptions of self, others, and personal agency assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in perceptions of self, others, and personal agency assessed using the Self-Descriptive Narrative and accompanying coding system as compared to baseline assessment.
Change from baseline in responsiveness in social interactions assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in responsiveness in social interactions assessed using the Social Responsiveness Scale as compared to baseline assessment. Higher scores are associated with greater responsiveness in social interactions
Change from baseline in sense of causation and personal agency assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in sense of causation and personal agency assessed using the Tones, Action Primes, and Agency Task as compared to baseline assessment.
Change from baseline in Big-5 personality traits assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in Big-5 personality traits assessed using the Ten-Item Personality Inventory as compared to baseline assessment. Higher scores are indicative of greater predilection to a specific Big 5 personality trait
Change from baseline in treatment motivation assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in treatment motivation assessed using the Treatment Motivation Questionnaire as compared to baseline assessment. Higher scores are indicative of greater treatment motivation
Change from baseline in loneliness assessed every six months for up to 24 months | Assessed at baseline and every six months throughout the completion of the study for up to 24 months
  Change in loneliness assessed using the UCLA Loneliness Scale as compared to baseline assessment. Higher scores are indicative of greater loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Breitborde, PhD, Principal Investigator — Ohio State University
Locations (1):
- OSU Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breitborde NJK, Guirgis H, Stearns W, Carpenter KM, Lteif G, Pine JG, Storey N, Wastler H, Moe AM. The Ohio State University Early Psychosis Intervention Center (EPICENTER) step-based care programme for individuals at clinical high risk for psychosis: study protocol for an observational study. BMJ Open. 2020 Jan 27;10(1):e034031. doi: 10.1136/bmjopen-2019-034031. PMID 31992606